CLINICAL TRIAL: NCT06947135
Title: The Effect of Targeted Stellate Ganglion Morphine Infiltration on Reperfusion Injury in STEMI Patients After Primary PCI: A Randomized Controlled Trial
Brief Title: Stellate Ganglion Morphine Infiltration on Myocardial Ischemia-Reperfusion Injury
Acronym: tSGM-AMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Ye Zhang, Senior doctor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YX2025-048
Record Dates: First submitted 2025-04-12; First posted 2025-04-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Stellate Ganglion; Percutaneous Coronary Intervention; Ischemia/reperfusion injury; Morphine
MeSH Terms: conditions — Reperfusion Injury | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine group (Experimental): Patients in the morphine group will receive a single injection of morphine (10 mg, 10 ml) around the left stellate ganglion under ultrasound guidance before coronary artery recanalization.
  Interventions: Drug: Morphine
- Saline group (Placebo Comparator): Patients in the placebo group will receive a single injection of 0.9% saline (10 ml) around the left stellate ganglion under ultrasound guidance before coronary artery recanalization.
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: Morphine — Morphine (10 mg, 10 ml) is injected around the stellate ganglion using ultrasound guidance prior to coronary artery recanalization
  Arms: Morphine group
Drug: saline placebo — Saline (10 ml) is injected around the stellate ganglion using ultrasound guidance prior to coronary artery recanalization
  Arms: Saline group

SUMMARY:
The goal of this clinical trial is to investigate whether morphine modulates the functions of the stellate ganglion to reduce myocardial ischemia/reperfusion injury in AMI patients. It will also assess the safety of injecting morphine around the stellate ganglion via ultrasound guidance. The main questions it aims to answer are:

1. Does morphine regulate stellate ganglion function to reduce myocardial ischemia/reperfusion injury in AMI patients?
2. What medical problems do participants experience when receiving injected morphine around the stellate ganglion? Researchers will compare morphine to a placebo saline (as a control group) to determine whether stellate ganglion infiltration with morphine effectively treats patients with AMI following primary PCI.

Participants will:

* Receive a single injection of morphine or saline around the stellate ganglion.
* Evaluate the percentage of infarct size 7 days after surgery, or at discharge if the duration is shorter than 7 days.
* Record their symptoms and any major adverse cardiovascular and cerebrovascular events within 30 days post-surgery.

DETAILED DESCRIPTION:
Acute ST-segment elevation myocardial infarction (STEMI) patients (aged ≥18 years) planned for percutaneous coronary intervention (PCI) will be enrolled for this study. Patients with severe complications of myocardial infarction, such as uncontrollable acute left heart failure or pulmonary edema, severe cardiogenic shock after cardiopulmonary resuscitation, severe mechanical complications including ventricular septal defect, papillary muscle rupture, and rupture of the left ventricular free wall; with old myocardial infarction, or cardiomyopathy, or malignant arrhythmias controlled by antiarrhythmic drugs; with coagulation disorders due to systemic diseases and those who are currently using anticoagulants and are not suitable for injection; with allergy to opioids or with a history of opioid addiction and those participating in other clinical studies; with pregnant or breastfeeding women; with severe organ dysfunction or failure; with severe infections; with severe mental illness that cannot cooperate and those taking antipsychotic drugs or considered unsuitable for this study by the researchers will be excluded. Subjects will be randomly assigned to one of two groups: the placebo group and the morphine group. Patients in the morphine group will receive a single injection of morphine (10 mg, 10 ml) around the left stellate ganglion under ultrasound guidance before coronary artery recanalization. Moreover, the placebo group will receive a 10 ml 0.9% saline infiltration around the stellate ganglion. The percentage of myocardial infarct size is measured by MRI either 7 days after primary PCI or at discharge if the duration is shorter than 7 days as the primary outcome. The secondary outcomes include the rate of major adverse cardiovascular and cerebrovascular events, cardiac function, rehospitalization rate, and mortality within 30 days; evaluation of myocardial injury during hospitalization, including cTnI levels and ECG examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, Male or Female.
2. Acute ST-segment elevation myocardial infarction (STEMI) patients planned for percutaneous coronary intervention (PCI). Acute STEMI is defined as: electrocardiogram shows ST-segment elevation ≥0.2 mV in two or more adjacent leads, or new left bundle branch block (LBBW).
3. Within 24 hours of the onset of infarct-related chest pain.
4. Obtaining informed consent from the patient and their family.

Exclusion Criteria:

1. Patients with severe complications of myocardial infarction, such as uncontrollable acute left heart failure and pulmonary edema, severe cardiogenic shock after cardiopulmonary resuscitation, severe mechanical complications including ventricular septal defect, papillary muscle rupture, and rupture of the left ventricular free wall;
2. Patients with old myocardial infarction, or cardiomyopathy, or malignant arrhythmias controlled by antiarrhythmic drugs;
3. Patients with coagulation disorders due to systemic diseases and those who are currently using anticoagulants and are not suitable for injection;
4. Patients allergic to opioids or with a history of opioid addiction and those participating in other clinical studies;
5. Pregnant or breastfeeding women;
6. Patients with severe organ dysfunction or failure, such as liver failure, renal failure, and respiratory failure;
7. Patients with severe infections;
8. Patients with severe mental illness that cannot cooperate and those taking antipsychotic drugs;
9. Other patients considered unsuitable for this study by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of myocardial infarct size | 7 days after primary PCI or at discharge
  The percentage of myocardial infarct size is measured by MRI either 7 days after primary PCI or at discharge if the duration is shorter than 7 days.

SECONDARY OUTCOMES:
The incidence of major adverse cardiovascular and cerebrovascular events (MACCE) | within 30 days post-surgery
  The incidence of MACCE, including cardiac death, rehospitalization for heart failure, recurrent myocardial infarction, coronary revascularization, and stroke, will be recorded within 30 days post-surgery.
Postoperative plasma hs-cTnI levels | at 24 hours post-surgery
  The levels of plasma hs-cTnI will be recorded at 24 hours post-surgery.
Evaluation of no-reflow phenomenon | at 2 hours, 24 hours or 7-day reperfusion
  The ST segment resolution will be evaluated by electrocardiograph (ECG) at 2 hours, 24 hours or 7-day reperfusion.
The incidence of microvascular obstruction | 7 days after primary PCI or at discharge
  The incidence of microvascular obstruction is evaluated by MRI either 7 days after primary PCI or at discharge if the duration is shorter than 7 days.
Major STEMI-related complications within 30 days post-surgery | within 30 days post-surgery
  The major STEMI-related complications, including cardiogenic shock, acute left heart failure, mechanical complications, malignant arrhythmias, will be recorded within 30 days post-surgery.
Rehospitalization rate due to cardiovascular adverse events | within 30 days post-surgery
  The rehospitalization rate due to cardiovascular adverse events will be recorded within 30 days post-surgery.
All-cause mortality | within 30 days post-surgery
  All-cause mortality will be recorded within 30 days post-surgery.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No